CLINICAL TRIAL: NCT00992589
Title: A Multi-Center, Double-Blind, Randomized, Placebo-Controlled, Parallel Group, Withdrawal Study to Evaluate the Safety and Efficacy of Delayed Release Rabeprazole in 1- to 11-Month-Old Pediatric Subjects With Symptomatic/Gastroesophageal Erosive Reflux Disease (GERD)
Brief Title: Safety and Efficacy of Rabeprazole in Infants With Gastroesophageal Erosive Reflux Disease (GERD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR014836; RABGRD3004 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2009-09-04; First posted 2009-10-09 (Estimated); Results first posted 2013-05-22 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-04

CONDITIONS: Gastroesophageal Reflux
Keywords: Gastroesophageal Reflux; Gastroesophageal Reflux Disease; GERD; Proton Pump Inhibitor; PPI; Regurgitation; Infants; AcipHex, PARIET; ALFENCE
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Rabeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rabeprazole sodium 5 mg (Experimental)
  Interventions: Drug: Rabeprazole sodium 5 mg
- Rabeprazole sodium 10 mg (Experimental)
  Interventions: Drug: Rabeprazole sodium 10 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rabeprazole sodium 5 mg — Rabeprazole Sodium 5 mg capsules once daily in the morning.
  Arms: Rabeprazole sodium 5 mg
Drug: Rabeprazole sodium 10 mg — Rabeprazole Sodium 10 mg capsules once daily in the morning.
  Arms: Rabeprazole sodium 10 mg
Drug: Placebo — Matching placebo capsules once daily in the morning.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effectiveness and safety of rabeprazole sodium, an inhibitor of gastric acid secretion of the protein pump inhibitor (PPI) class, compared with placebo in the treatment of gastrointestinal esophageal reflux disease (GERD) in infants 1 to 11 months of age.

DETAILED DESCRIPTION:
Rabeprazole sodium belongs to the class of drugs known as proton pump inhibitors, which suppress gastric acid secretion. The drug is approved in the United States for the treatment of adults with GERD and other acid-related gastrointestinal disorders, and has been studied in adolescents (older than 12 years of age) with results similar to those in adults. However, the drug has not been studied in children under the age of 12 years. This study focuses on the efficacy and safety of rabeprazole sodium in infants aged 1 to 11 months, the pediatric group in which the prevalence of GERD-related symptoms is the greatest. This is a multicenter, double-blind, randomized, placebo-controlled, parallel-group withdrawal study to compare the efficacy and safety of 2 doses (0.5 mg/kg or 1.0 mg/kg daily) of rabeprazole with placebo in the treatment of infants aged 1 to 11 months who have a diagnosis of suspected GERD, symptomatic GERD, or endoscopically or histologically proven GERD. The study consists of 3 study periods: a screening period of up to 10 days, an open-label treatment period of up to 3 weeks, and a 5-week double-blind treatment period. Patients who have been receiving GERD therapy before screening will have their GERD therapy discontinued for 3 days before entering the open-label treatment period. Patients who have a positive clinical response according to the Clinical Global Impressions - Improvement (CGI-I) scale at the end of the first or second week of the open-label treatment period will enter the double-blind treatment period; those who do not will be withdrawn from the study. A parent, legal guardian, or other individual experienced in the care of the infant will be the primary caregiver, who is responsible for the daily and weekly assessments and study drug administration. Efficacy assessments consist of the Infant Gastroesophageal Reflux Questionnaire Revised (I GERQ-R) total score, the Infant Gastroesophageal Reflux Questionnaire-Daily Diary (I GERQ-DD) total score, the CGI-I, the Global Treatment Satisfaction Score, and the weight-for-age Z-score. Safety assessments include monitoring of concomitant therapies and adverse events throughout the study; clinical laboratory testing (hematology, clinical chemistry, urinalysis), measurement of vital signs (pulse and respiratory rate, blood pressure, temperature); and physical examination including length and weight. The study hypothesis is that rabeprazole sodium is superior to placebo in the treatment of GERD in infants aged 1 to 11 months. Rabeprazole sodium capsule(s) by mouth once a day, 10.0 milligram (mg)/kilogram (kg) for up to 3 weeks during the open-label treatment period and either 5.0 mg/kg or 10.0 mg/kg during the 5-week double-blind treatment period. To give the study drug to the infants, the contents of the capsule(s) are sprinkled onto a small amount of soft food or, as needed, the contents of the capsule(s) may be given in a small amount (5 milliliter [mL]) of infant formula or expressed breast milk.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of suspected GERD, symptomatic GERD, or endoscopically or histologically proven GERD, based on frequent vomiting or regurgitation, with at least 1 of the following: a) poor weight gain, or b) irritability, excessive crying or disturbed sleep that both the parent(s) and the doctor consider abnormal (but not due to colic)
* or c) refusal to eat even if hungry or arching of the back during meals
* weight 2.5 kg to 15.0 kg
* I-GERQ-R score >16
* Have only 1 caregiver in addition to the parent(s)

Exclusion Criteria:

* History of confirmed acute life-threatening events due to GERD
* Known narrowing of the opening from the stomach to the small intestines
* Confirmed diagnosis of cow's milk allergy
* Have taken PPIs or H2-blockers (a class of drugs that inhibit stomach acid production) or any of several drugs that affect the normal movement of the digestive tract (caffeine, theophylline, antacids, erythromycin, and others) within 3 days before entering the study
* Have blood or urine test results that are well above or below the normal range for the infant

Ages: 1 Month to 11 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 344 (Actual)
Dates: Start 2009-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (81):
- United States (43):
  - Birmingham, Alabama
  - Columbiana, Alabama
  - Dothan, Alabama
  - Huntsville, Alabama
  - Mobile, Alabama
  - Phoenix, Arizona
  - Bentonville, Arkansas
  - Orange, California
  - Centennial, Colorado
  - Thornton, Colorado
  - Maitland, Florida
  - Miami, Florida
  - Augusta, Georgia
  - Park Ridge, Illinois
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - Owensboro, Kentucky
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Flint, Michigan
  - Saint Paul, Minnesota
  - Jackson, Mississippi
  - Bridgeton, Missouri
  - Mays Landing, New Jersey
  - Valhalla, New Jersey
  - Buffalo, New York
  - The Bronx, New York
  - Utica, New York
  - Charlotte, North Carolina
  - Toledo, Ohio
  - Youngstown, Ohio
  - Gresham, Oregon
  - Hershey, Pennsylvania
  - Chattanooga, Tennessee
  - Kingsport, Tennessee
  - Dallas, Texas
  - Laredo, Texas
  - San Antonio, Texas
  - Tomball, Texas
  - Fairfax, Virginia
  - Huntington, West Virginia
- Australia (5):
  - Garran
  - Herston
  - Kogarah
  - Parkville
  - Sydney
- Belgium (3):
  - Antwerp
  - Brussels
  - Leuven
- Pleven, Bulgaria
- Odense, Denmark
- Hungary (9):
  - Békéscsaba
  - Budapest
  - Gyõr
  - Gyulai Ut 18
  - Miskolc
  - Nyíregyháza
  - Pécs
  - Szombathely
  - Veszprém
- Israel (6):
  - Haifa
  - Jerusalem
  - Petach Tikvah
  - Petah Tikva
  - Ramat Gan
  - Tiberias
- Netherlands (3):
  - Amsterdam
  - Nijmegen
  - Zwolle
- Poland (6):
  - Bialystok
  - Bydgoszcz
  - Częstochowa
  - Rzeszów
  - Torun
  - Warsaw
- South Africa (4):
  - Durban
  - Durbanville
  - Panorama
  - Wynberg

REFERENCES:
- [Derived] Sharp WG, Stubbs KH, Adams H, Wells BM, Lesack RS, Criado KK, Simon EL, McCracken CE, West LL, Scahill LD. Intensive, Manual-based Intervention for Pediatric Feeding Disorders: Results From a Randomized Pilot Trial. J Pediatr Gastroenterol Nutr. 2016 Apr;62(4):658-63. doi: 10.1097/MPG.0000000000001043. PMID 26628445
- [Derived] Hussain S, Kierkus J, Hu P, Hoffman D, Lekich R, Sloan S, Treem W. Safety and efficacy of delayed release rabeprazole in 1- to 11-month-old infants with symptomatic GERD. J Pediatr Gastroenterol Nutr. 2014 Feb;58(2):226-36. doi: 10.1097/MPG.0000000000000195. PMID 24121146
- [Derived] Treem W, Hu P, Sloan S. Normal and proton pump inhibitor-mediated gastrin levels in infants 1 to 11 months old. J Pediatr Gastroenterol Nutr. 2013 Oct;57(4):520-6. doi: 10.1097/MPG.0b013e31829b6914. PMID 23689261

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-Label Rabeprazole Sodium 10 mg; Double-Blind Rabeprazole Sodium 5 mg; Double-Blind Rabeprazole Sodium 10 mg: Rabeprazole Sodium capsules once daily in the morning.
- Double-Blind Placebo: Matching placebo capsules once daily in the morning.
Period: Open-Label Phase
Arm/Group | Open-Label Rabeprazole Sodium 10 mg | Double-Blind Placebo | Double-Blind Rabeprazole Sodium 5 mg | Double-Blind Rabeprazole Sodium 10 mg
Started | 344 | 0 | 0 | 0
Completed | 267 | 0 | 0 | 0
Not Completed | 77 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 20 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 3 | 0 | 0 | 0
Not completed — Physician Decision | 4 | 0 | 0 | 0
Not completed — Other | 45 | 0 | 0 | 0
Period: Double-Blind Phase
Arm/Group | Open-Label Rabeprazole Sodium 10 mg | Double-Blind Placebo | Double-Blind Rabeprazole Sodium 5 mg | Double-Blind Rabeprazole Sodium 10 mg
Started | 0 | 89 | 90 | 88
Completed | 0 | 76 | 77 | 78
Not Completed | 0 | 13 | 13 | 10
Not completed — Adverse Event | 0 | 6 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 6 | 5 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2
Not completed — Other | 0 | 1 | 6 | 3

BASELINE CHARACTERISTICS:
Arm/Group | Open-Label Rabeprazole Sodium 10 mg
Number analyzed (Participants) | 344
Age Continuous [Mean (Standard Deviation); unit: months] | 4.6 (2.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139
  Male | 205
Region of Enrollment [Number; unit: participants]
  AUSTRALIA | 7
  BELGIUM | 11
  BULGARIA | 24
  HUNGARY | 51
  ISRAEL | 36
  ITALY | 5
  NETHERLANDS | 9
  POLAND | 56
  SOUTH AFRICA | 12
  UNITED STATES | 133
AgeCategorical [Number; unit: participants]
  >= 1 to < 4 Months | 175
  >= 4 to < 8 Months | 124
  >= 8 to < 12 Months | 45

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Daily Frequency of Regurgitation (Double-blind Phase/ Baseline Observation Carried Forward)
Time Frame: Baseline, Week 8
Population: Intent to Treat population, which consisted of all participants who completed the Open-label period, were randomly assigned to treatment in the Double-blind (DB) period, had taken at least 1 dose of DB study drug, and with evaluable data at each measurement time point.
Measure: Mean (Standard Deviation); unit: frequency of Regurgitation
Groups:
- Double-Blind Rabeprazole Sodium Total: Rabeprazole Sodium capsules once daily in the morning.
Arm/Group | Double-Blind Placebo | Double-Blind Rabeprazole Sodium 5 mg | Double-Blind Rabeprazole Sodium 10 mg | Double-Blind Rabeprazole Sodium Total
Number analyzed (Participants) | 88 | 88 | 85 | 173
frequency of Regurgitation | -0.8 (1.58) | -0.8 (1.55) | -1.6 (3.63) | -1.2 (2.79)
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Rabeprazole Sodium Total; Analysis of Covariance with Treatment as fixed effect, Region and Age as stratification factors and Change from Open-label (OL) Baseline to OL Endpoint as covariate to test the hypothesis of no difference in change in daily average frequency of regurgitation from Double-blind (DB) Baseline to DB Endpoint between rabeprazole sodium total and placebo; Test type: Superiority or Other; p = 0.168, ANCOVA; Least-Squares Mean Difference = -0.449, 95% CI 2-sided [-1.087 to 0.190]

2. Primary Outcome: Change From Baseline in Weight-for-Age Z-Score (Double-blind Phase/ Baseline Observation Carried Forward)
Description: Body weight was measured with the participant unclothed and before a feeding during each office visit. In the analysis of weight data, weight will be transformed to the weight-for-age Z-score using World Health Organization Child Growth Standards, taking into account the infant's age and gender (Borghi E, 2006).
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Double-Blind Placebo | Double-Blind Rabeprazole Sodium 5 mg | Double-Blind Rabeprazole Sodium 10 mg | Double-Blind Rabeprazole Sodium Total
Number analyzed (Participants) | 89 | 90 | 88 | 178
Z-score | 0.11 (0.329) | 0.16 (0.322) | 0.11 (0.264) | 0.14 (0.295)
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Rabeprazole Sodium Total; Analysis of Covariance with Treatment as fixed effect, Region and Age as stratification factors and Double-blind (DB) Baseline as covariate to test the hypothesis of no difference in change in Weight-for-Age Z-Score from DB Baseline to DB Endpoint between Rabeprazole Sodium Total and Placebo; Test type: Superiority or Other; p = 0.440, ANCOVA; Least-Squares Mean Difference = 0.030, 95% CI 2-sided [-0.047 to 0.108]

3. Secondary Outcome: The Daily Average Number of Episodes Related to Each Volume of Regurgitation During the Double-blind Treatment Period
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of episodes
Groups:
- Double-Blind Placebo - Baseline; Double-Blind Placebo - Week 8: Matching placebo capsules once daily in the morning.
- Double-Blind Rabeprazole Sodium 5 mg - Baseline; Double-Blind Rabeprazole Sodium 10 mg - Baseline; Double-Blind Rabeprazole Sodium 5 mg - Week 8; Double-Blind Rabeprazole Sodium 10 mg - Week 8; Double-Blind Rabeprazole Sodium Total - Baseline; Double-Blind Rabeprazole Sodium Total - Week 8: Rabeprazole Sodium capsules once daily in the morning.
Arm/Group | Double-Blind Placebo - Baseline | Double-Blind Rabeprazole Sodium 5 mg - Baseline | Double-Blind Rabeprazole Sodium 10 mg - Baseline | Double-Blind Placebo - Week 8 | Double-Blind Rabeprazole Sodium 5 mg - Week 8 | Double-Blind Rabeprazole Sodium 10 mg - Week 8 | Double-Blind Rabeprazole Sodium Total - Baseline | Double-Blind Rabeprazole Sodium Total - Week 8
Number analyzed (Participants) | 89 | 90 | 88 | 89 | 90 | 88 | 178 | 178
number of episodes
  Less than 1 tablespoon | 1.2 (2.52) | 1.1 (1.49) | 1.9 (4.25) | 0.8 (2.15) | 0.7 (1.35) | 1.0 (1.92) | 1.5 (3.18) | 0.9 (1.66)
  1 to 2 tablespoons | 0.7 (1.04) | 0.7 (1.08) | 1.2 (1.73) | 0.5 (1.62) | 0.4 (0.75) | 0.7 (1.55) | 1.0 (1.45) | 0.6 (1.21)
  More than 2 tablespoons to 2 fluid oz | 0.3 (0.53) | 0.2 (0.43) | 0.3 (0.77) | 0.2 (0.48) | 0.1 (0.60) | 0.2 (0.65) | 0.2 (0.62) | 0.2 (0.63)
  More than 2 fluid oz to 4 fluid oz | 0.1 (0.19) | 0.0 (0.09) | 0.0 (0.08) | 0.0 (0.09) | 0.0 (0.14) | 0.0 (0.23) | 0.0 (0.08) | 0.0 (0.19)
  More than 4 fluid oz | 0.0 (0.05) | 0.0 (0.14) | 0.0 (0.24) | 0.0 (0.11) | 0.0 (0.05) | 0.0 (0.04) | 0.0 (0.20) | 0.0 (0.04)

4. Secondary Outcome: Change From Baseline in Weekly Average I-GERQ-DD Regurgitation Subscale Score (Double-blind Phase/ Last Observation Carried Forward)
Description: The Infant Gastroesophageal Reflux Questionnaire-Daily Diary (I-GERQ-DD) is a 9-item daily diary that the primary caregiver will be instructed to complete every evening at the same time interval after the participant has gone to sleep for the night. The I-GERQ-DD contains 3 subscales: the Regurgitation subscale, the Eating Behavior subscale and the Discomfort subscale. The Regurgitation subscale will be calculated as the sum of the 3 questions regarding regurgitation (Questions 1, 2, 3) and will range from 0 to 13. For each subscale score, a higher value indicates a worse outcome.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Double-Blind Placebo | Double-Blind Rabeprazole Sodium 5 mg | Double-Blind Rabeprazole Sodium 10 mg | Double-Blind Rabeprazole Sodium Total
Number analyzed (Participants) | 88 | 88 | 85 | 173
scores on a scale | -0.8 (2.57) | -0.8 (2.56) | -1.0 (2.38) | -0.9 (2.47)
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Rabeprazole Sodium Total; Analysis of Covariance with Treatment as fixed effect, Region and Age as stratification factors and Change from Open-label (OL) Baseline to OL Endpoint as covariate to test the hypothesis of no difference in change in weekly average I-GERQ-DD Regurgitation Subscale Score from Double-blind (DB) Baseline to DB Endpoint between rabeprazole sodium total and placebo; Test type: Superiority or Other; p = 0.984, ANCOVA; Least-Squares Mean Difference = 0.006, 95% CI 2-sided [-0.619 to 0.632]

5. Secondary Outcome: Change From Baseline in Weekly Average I-GERQ-DD Discomfort Subscale Score (Double-blind Phase/ Last Observation Carried Forward)
Description: The Infant Gastroesophageal Reflux Questionnaire-Daily Diary (I-GERQ-DD) is a 9-item daily diary that the primary caregiver will be instructed to complete every evening at the same time interval after the subject has gone to sleep for the night. The I-GERQ-DD contains 3 subscales: the Regurgitation subscale, the Eating Behavior subscale and the Discomfort subscale. The Discomfort subscale score will be calculated as the sum of the 3 questions regarding discomfort (Questions, 7, 8, 9) and will range from 0 to 12. For each subscale score, a higher value indicates a worse outcome.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Double-Blind Placebo | Double-Blind Rabeprazole Sodium 5 mg | Double-Blind Rabeprazole Sodium 10 mg | Double-Blind Rabeprazole Sodium Total
Number analyzed (Participants) | 88 | 88 | 85 | 173
scores on a scale | 0.0 (2.24) | -0.1 (1.88) | -0.4 (1.94) | -0.2 (1.9)
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Rabeprazole Sodium Total; Analysis of Covariance with Treatment as fixed effect, Region and Age as stratification factors and Change from Open-label (OL) Baseline to OL Endpoint as covariate to test the hypothesis of no difference in change in weekly average I-GERQ-DD Discomfort Subscale Score from Double-blind (DB) Baseline to DB Endpoint between rabeprazole sodium total and placebo; Test type: Superiority or Other; p = 0.479, ANCOVA; Least-Squares Mean Difference = -0.182, 95% CI 2-sided [-0.690 to 0.325]

6. Secondary Outcome: Change From Baseline in Weekly Average I-GERQ-DD Eating Behavior Subscale Score (Double-blind Phase/ Last Observation Carried Forward)
Description: The Infant Gastroesophageal Reflux Questionnaire-Daily Diary (I-GERQ-DD) is a 9-item daily diary that the primary caregiver will be instructed to complete every evening at the same time interval after the subject has gone to sleep for the night. The I-GERQ-DD contains 3 subscales: the Regurgitation subscale, the Eating Behavior subscale and the Discomfort subscale. The Eating Behavior subscale score will be calculated as the sum of the 3 questions regarding eating behavior (Questions 4, 5, 6) and will range from 0 to 12. For each subscale score, a higher value indicates a worse outcome.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Double-Blind Placebo | Double-Blind Rabeprazole Sodium 5 mg | Double-Blind Rabeprazole Sodium 10 mg | Double-Blind Rabeprazole Sodium Total
Number analyzed (Participants) | 88 | 88 | 85 | 173
scores on a scale | -0.1 (2.54) | -0.1 (2.19) | -0.4 (2.15) | -0.3 (2.17)
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Rabeprazole Sodium Total; Analysis of Covariance with Treatment as fixed effect, Region and Age as stratification factors and Change from Open-label (OL) Baseline to OL Endpoint as covariate to test the hypothesis of no difference in change in weekly average I-GERQ-DD Eating Behavior Subscale Score from Double-blind (DB) Baseline to DB Endpoint between rabeprazole sodium total and placebo; Test type: Superiority or Other; p = 0.498, ANCOVA; Least-Squares Mean Difference = -0.192, 95% CI 2-sided [-0.751 to 0.366]

7. Primary Outcome: Change From Baseline in I-GERQ-R Total Score (Double-blind Phase/ Baseline Observation Carried Forward)
Description: The Infant Gastroesophageal Reflux Questionnaire-Revised (I-GERQ-R) is a 12-item questionnaire that is completed by the primary caregiver at every office or telephonic visit. It has a weekly recall and the items cover the frequency, amount and discomfort attributed to spit-up, refusal or stopping feeding, crying and fussing, hiccups, arching back and stopping breathing or changing color. The total score is calculated as the sum of all 12 scores for the individual questions, and ranges from 0 to 42. A higher value indicates a worse outcome.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Double-Blind Placebo | Double-Blind Rabeprazole Sodium 5 mg | Double-Blind Rabeprazole Sodium 10 mg | Double-Blind Rabeprazole Sodium Total
Number analyzed (Participants) | 89 | 89 | 87 | 176
scores on a scale | -3.6 (6.41) | -3.8 (7.5) | -4.1 (7) | -3.9 (7.24)
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Rabeprazole Sodium Total; Analysis of Covariance with Treatment as fixed effect, Region and Age as stratification factors and Change from Open-label (OL) Baseline to OL Endpoint as covariate to test the hypothesis of no difference in change in I-GERQ-R Total Score from Double-blind (DB) Baseline to DB Endpoint between rabeprazole sodium total and placebo; Test type: Superiority or Other; p = 0.960, ANCOVA; Least-Squares Mean Difference = 0.042, 95% CI 2-sided [-1.615 to 1.700]

8. Primary Outcome: Change From Baseline in in Weekly Average I-GERQ-DD Total Score (Double-blind Phase/ Baseline Observation Carried Forward)
Description: The Infant Gastroesophageal Reflux Questionnaire-Daily Diary (I-GERQ-DD) is a 9-item daily diary that the primary caregiver will be instructed to complete every evening at the same time interval after the participant has gone to sleep for the night. The I-GERQ-DD contains 3 subscales: the Regurgitation subscale, the Eating Behavior subscale and the Discomfort subscale. Each of the 9 items will be assigned a numeric score. The total score will be calculated as the sum of all 9 items, and ranges from 0 to 37. A higher value indicates a worse outcome.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Double-Blind Placebo | Double-Blind Rabeprazole Sodium 5 mg | Double-Blind Rabeprazole Sodium 10 mg | Double-Blind Rabeprazole Sodium Total
Number analyzed (Participants) | 88 | 88 | 85 | 173
scores on a scale | -1.9 (4.55) | -1.6 (4.85) | -2.1 (4.9) | -1.9 (4.86)
Statistical Analysis 1: Comparison: Double-Blind Placebo vs Double-Blind Rabeprazole Sodium Total; Analysis of Covariance with Treatment as fixed effect, Region and Age as stratification factors and Change from Open-label (OL) Baseline to OL Endpoint as covariate to test the hypothesis of no difference in change in Weekly Average I-GERQ-DD Total Score from Double-blind (DB) Baseline to DB Endpoint between rabeprazole sodium total and placebo; Test type: Superiority or Other; p = 0.968, ANCOVA; Least-Squares Mean Difference = 0.024, 95% CI 2-sided [-1.167 to 1.214]

ADVERSE EVENTS:
Arm/Group | Open-Label Rabeprazole Sodium 10 mg | Double-Blind Placebo | Double-Blind Rabeprazole Sodium 5 mg | Double-Blind Rabeprazole Sodium 10 mg
Serious Adverse Events (participants affected / at risk) | 15/344 | 2/89 | 8/90 | 3/88
Other Adverse Events (participants affected / at risk) | 116/344 | 33/89 | 34/90 | 32/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label Rabeprazole Sodium 10 mg (N=344) | Double-Blind Placebo (N=89) | Double-Blind Rabeprazole Sodium 5 mg (N=90) | Double-Blind Rabeprazole Sodium 10 mg (N=88)
Hypoacusis (Ear and labyrinth disorders) | 1 | 1 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 0 | 2 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 0 | 2 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 0 | 2 | 0
Viral Infection (Infections and infestations) | 1 | 0 | 0 | 1
Beta 2 Microglobulin Increased (Investigations) | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Failure to Thrive (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 1 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label Rabeprazole Sodium 10 mg (N=344) | Double-Blind Placebo (N=89) | Double-Blind Rabeprazole Sodium 5 mg (N=90) | Double-Blind Rabeprazole Sodium 10 mg (N=88)
Constipation (Gastrointestinal disorders) | 15 | 4 | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 21 | 7 | 8 | 4
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 13 | 7 | 2 | 4
Vomiting (Gastrointestinal disorders) | 13 | 5 | 6 | 2
Pyrexia (General disorders) | 22 | 5 | 9 | 6
Nasopharyngitis (Infections and infestations) | 19 | 4 | 8 | 3
Otitis Media (Infections and infestations) | 14 | 4 | 5 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 19 | 6 | 3 | 8
Blood Gastrin Increased (Investigations) | 10 | 0 | 2 | 7
Rash (Skin and subcutaneous tissue disorders) | 12 | 4 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less